CLINICAL TRIAL: NCT07259499
Title: Towards an Integrated Care System for the Assistance of Patients With Chronic Diseases, Multimorbidity, Frailty, and Polypharmacy
Brief Title: Predictors of Emergency Department Use in Frail Patients
Acronym: THE-Spoke 10
Status: Recruiting | Type: Observational
Sponsor: University of Pisa (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Gabriele Siciliano, Professor, MD, PhD, University of Pisa
Other Study IDs: 25312_SICILIANO
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer s Disease; Vascular Dementia; Frailty; Elderly; Emergency Department Visits; Autonomy
Keywords: phosphorylated tau 181; dementia; Emergency Department; Frailty; Autonomies; Elderly; cerebrovascular
MeSH Terms: conditions — Dementia, Vascular; Frailty; Dementia; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly, non-autonomous Patients: Adult participants fulfilling the following inclusion criteria: fluency in Italian language, age higher than 64 years, loss of autonomies of daily living as assessed by the Katz Activities of Daily Living or in the Lawton Instrumental Activities of Daily Living questionnaires, having performed blood exams and a head neuroimaging feasable for cerebrovascular burden assessment, i.e., Magnetic Resonance Imaging (MRI) or computed tomography (CT), in the 6 months prior to recruitment.
  Interventions: Diagnostic Test: Plasma phosphorylated Tau 181

INTERVENTIONS:
Diagnostic Test: Plasma phosphorylated Tau 181 — Plasma will be collected in dipotassium EDTA tubes at recruitment and centrifugated at 1800-2000xg for 10 minutes within a short data frame. Plasma will be subsequently aliquoted and stored at -80°C. Immediately prior to analysis, samples will be thawed at room temperature, vortexed, and centrifuged. Plasma p-tau181 concentrations will be then quantified using a fully automated chemiluminescent enzyme immunoassay on the LUMIPULSE G600II system, in accordance with the manufacturer's instructions.

SUMMARY:
When admitted to the emergency department (ED), elderly non-autonomous patients show high risk of adverse health outcomes. The prompt identification of ED use risk factors in such population is hence needed. While cognitive impairment is a known clinical risk factor, biomarkers of most prevalent dementias have been scarcely investigated as possible ED use predictors. Within this context, this prospective study aims at exploring whether plasma phospho-tau181 and cerebrovascular burden can predict ED use at 6 months in elderly non-autonomous patients, irrespective of frailty.

DETAILED DESCRIPTION:
When admitted to the emergency department (ED), elderly non-autonomous patients show high risk of mortality, extended hospital stays and early readmission after discharge. The prompt identification of ED use risk factors in such population is hence urgently needed. Among these, cognitive impairment emerged as a key neurologic risk factor of ED use.

Alzheimer's Disease (AD) and cerebrovascular damage are the first cause of cognitive impairment in the general population. Several biomarkers have been proposed to distinguish different types of dementia during clinical practice. Considering AD, plasma phosphorylated tau 181 protein (ptau181) recently emerged as a biomarker which accurately predicts cerebrospinal ptau181 levels. Moreover, based on this evidence and on its minimally invasive nature, plasma ptau181 has been recently proposed as a biomarker to be employed during the AD diagnostic process, along with previously recommended procedures. Of note, plasma pTau181 levels are positively associated to confusional state risk in hospitalized patients. In parallel, cerebrovascular burden is commonly assessed in available neuroimages during the clinical characterization of cognitive impairments, and its severity has been associated to the severity of cognitive impairment. Within this context, no studies explored biomarkers of AD and vascular dementia as possible risk factors for ED use. Confirming such predictive value may result highly useful in stratifying the patients' risk of future adverse health outcomes during clinical practice.

Of note, non-autonomous elderly patients often suffer from multiple health problems. Such health problems concur to define patients' frailty, with higher frailty levels being associated with increased rates of adverse health outcomes, included ED use and mortality. Due to the multidimensional nature of frailty, several assessment methods have been developed. Specifically, recent literature proposed the use of multidimensional frailty indexes including relatively extended sets of variables available in public health databases. Among these, routinary assessed blood biomarkers and scales characterizing frailty from different clinical standpoints, e.g., nutritional status, autonomies of daily living, lower limb functionality, have been included. Demonstrating a relationship between biomarkers of cognitive impairment and ED use irrespective of patients' multidimensional frailty would highlight the importance of the neurological evaluation within the clinical assessment of non-autonomous elderly patients.

Within this context, the present study aims at investigating whether plasma ptau181 and cerebrovascular burden can predict ED use in non-autonomous elderly patients within a relatively short observational period, irrespective of multidimensional clinical frailty.

ELIGIBILITY:
Inclusion Criteria:

* fluency in Italian language,
* age higher than 64 years,
* loss of autonomies of daily living as assessed by the Katz Activities of Daily Living or in the Lawton Instrumental Activities of Daily Living questionnaires,
* having performed routinary blood exams in the 6 months prior to recruitment
* having performed head neuroimaging feasable for cerebrovascular burden assessment, i.e., Magnetic Resonance Imaging (MRI) or computed tomography (CT), in the 6 months prior to recruitment.

Exclusion Criteria:

* withdrawal of the informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults fulfilling the inclusion criteria consecutively recruited during their outpatient visits at the Neurology and Geriatrics Units of the Pisa University Hospital (Italy).
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-11-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Emergency Department Use | Within 6 months from recruitment
  The patient visits an emergency department (ED). The proportion of participants visiting the ED will be assessed at the end of the observational period.
  Biomarkers of cognitive impairment, i.e., plasma phosphorylated tau 181 and cerbrovascular burden, will be subsequently tested as possible predictors of this outcome.

SECONDARY OUTCOMES:
Time to emergency department use | Within 6 months from recruitment.
  The difference in days between the emergency department (ED) use and the recruitment date.
  The mean time to emergency department use will be assessed in ED users at the end of the observational period.
  Biomarkers of cognitive impairment, i.e., plasma phosphorylated tau 181 and cerbrovascular burden, will be subsequently tested as possible predictors of this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Siciliano, Professor, MD, PhD, Principal Investigator — University of Pisa
Locations (1):
- Azienda Ospedaliera Universitaria Pisana, Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication.
Access Criteria: The anonymized data underlying this article will be shared on reasonable request to the corresponding author of the published study.